CLINICAL TRIAL: NCT05960266
Title: Immunological Analysis of Lymph Node Tissue After Intralymphatic Immunotherapy: A Prospective Case Control Study
Acronym: ILIT-FNA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-00821
Record Dates: First submitted 2023-06-23; First posted 2023-07-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hypersensitivity; Hay Fever; Rhinitis, Allergic, Seasonal; Rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: One arm of patients will be treated by subcutaneous immunotherapy (SCIT). A second arm of patients will be treated by intralymphatic immunotherapy (ILIT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous immunotherapy (Active Comparator): Subcutaneous injection of grass-rye pollen allergen extract and micro-crystalline tyrosine.
  Single dose of 2000 U allergen in 0.5 ml. Dosage form: aqueous suspension.
  Interventions: Biological: Polvac Grass+Rye
- Intralymphatic immunotherapy (Experimental): Subcutaneous injection of grass-rye pollen allergen extract and micro-crystalline tyrosine.
  Single dose of 400 U allergen in 0.1 ml. Dosage form: aqueous suspension.
  Interventions: Biological: Polvac Grass+Rye

INTERVENTIONS:
Biological: Polvac Grass+Rye — Aqueous suspension of a co-precipitate of allergen extract and tyrosine

SUMMARY:
Allergy is a public health problem as more than 20% of western society is affected by it. Symptomatic treatment of allergy suffices with less severe allergy. Patients with more severe allergy should be treated with allergen immunotherapy (AIT). Present options of AIT are efficient but of long duration, associated with side effects and require much time from the patient. With Intralymphatic immunotherapy (ILIT), allergen is injected into the lymph node under ultrasound guidance. ILIT is complete after 3 treatment visits, may be more effective than and may have markedly fewer side effects than presently available methods of AIT.

The investigators plan a randomized, parallel group, open-label, prospective case-control study to assess immunological changes in lymph node and peripheral blood after intralymphatic (ILIT) or subcutaneous (SCIT) immunotherapy with POLVAC.

The intervention consists of one ultrasound-guided injection of allergen into inguinal lymph node or subcutaneous injection 1 cm next to the lymph node. Intervention quality (accuracy of injection) will be assessed by the administering physician during treatment and via video recording on the ultrasound device. Side effects associated with treatment will be recorded by the patients for 3 days after the injection.

The effect of intralymphatic or subcutaneous injection on lymph node tissue and immunoglobulins E and G4 in serum as well as cellular analyses of lymph node tissue and peripheral blood will be determined in samples taken during the trial.

The primary effect parameter is the effect of a single intralymphatic allergen injection on immunological parameters as well as allergen delivery to the lymph node as compared with a single subcutaneous injection.

DETAILED DESCRIPTION:
This is a prospective, comparative, clinical open label pilot study. From patients with grass pollen allergy who undergo a pre-seasonal SCIT scheme with Polvac™ Grass+RyeSCIT at the USZ Allergy Unit, 30 patients will be recruited for the study.

Four to six weeks after end of SCIT treatment (at maximal maintenance dose), the patients will be randomized to one out of two treatment groups and receive one additional allergen injection. Both treatment groups receives the same drug, but at different doses and routes of administration. Fifteen patients will be allocated to receive another subcutaneous injection with 0.5 ml (2000 U) Polvac Grass+Rye. The other 15 patients will be allocated to receive an intralymphatic injection of 0.1 ml Polvac Grass+Rye with 400 U allergen. Both SCIT and ILIT injections are performed by ultrasound-guidance as to assure injection into the lymph node (ILIT) or 1 cm next to the lymph node (SCIT).

The FNA of lymph node tissue will be conducted at 2, 6 or 24 hours after allergen injection. At the same time, FNA of a contralateral lymph nodes will be performed as baseline. Venous blood will be sampled at all visits: at baseline as well as after 2, 6 or 24 hours, after 7 days and after 28 days of the allergen ILIT or SCIT. The FNA is performed by ultrasound-guidance.

Drug preparation:

The 1 ml medication vial (4000 U/ml) is shaken for 10 seconds. The head of the vial is disinfected and 0.5 ml (for SCIT) or 0.1 ml (for ILIT) of the medication is drawn into a 1 ml syringe with 23G hypodermic needle assuring no air in the syringe or needle. The medication is used no later than 4 hours after the preparation. Replica of the dose are made if more than one injection is to be performed. The remaining medication is discarded.

Fine needle aspiration (FNA):

The FNA is minimally invasive and performed by an experienced investigator. The skin above the lymph node, will be disinfected and a sterile needle (23-25g), attached to the 5 ml syringe, fixed in a FNA gun, will be inserted into the lymph node cortex under colour Doppler ultrasound guidance while avoiding important tissues and organs, such as large blood vessels and nerves. The syringe plunger is drawn to set the seal at a 2 ml scale in order to maintain negative pressure in the syringe. After rotating and aspirating the syringe 5 times, the needle is rotated to aspirate in a fan shape way at different trajectories in the lymph node. The needle is withdrawn when ca. 0.1 ml tissue is present in the syringe. The puncture site is covered with sterile gauze and pressure is applied with appropriate force for 10 min. Patients are observed for 30 min of observation and released when no adverse reaction. The FNA sample will be rinsed with dimethyl sulfoxide (DMSO)-containing live cell freezing medium (10% DMSO and 90% fetal bovine serum (FBS)), put into a cryotube and frozen in -80°C.

Blood collection and preservation of cells and blood serum:

Venous blood collection is performed just before SCIT/ILIT, at 2, 6 or 24 hours post SCIT/ILIT, and at 7 and 28 post SCIT/SLIT. Each time, 25 ml venous blood is collected for preparation of PBMCs and 5 ml blood is collected for preparation of serum. Both samples are processed by routine in-house methods within 2 hours for preparation of serum and cells. The produced serum is aliquoted in 1 ml samples and frozen at - 20 °C for later analysis. Whole blood is centrifuged on Ficoll and the PBMCs isolated and washed in PBS before re-suspended in DMSO-containing live cell freezing medium. 1 ml aliquots of the cells are slow-frozen in cryotubes and finally stored at -80 °C before further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have seasonal grass-pollen-induced rhinoconjunctivitis as confirmed by patient history and type-1-sensitization to grass-pollen in skin and/or serum.
* Patients that undergo pre-seasonal short-term scheme with Polvac™ SCIT at the USZ Allergy Unit in autumn and winter 2023 for treatment of allergic rhinoconjunctivitis.

Informed Consent as documented by signature.

* Patients are between 18 and 55 years of age when they sign the informed consent.

Exclusion Criteria:

* Known or suspected allergy to additives to the study product
* Known intolerance or allergy to phenol
* Planned depot steroid injection for treatment of allergic rhinoconjunctivitis
* Uncontrolled asthma or severe asthma with post bronchodilator FEV1<70%, decided by the investigator
* Pulmonary disease with post bronchodilator FEV1 < 70 % of predicted
* Pulmonary disease, perennial or seasonal, with daily use of more than 800 microgram inhaled budesonide/day (or equivalent)
* Treatment with omalizumab or other biologics for allergy, AD, urticaria or asthma.
* Allergic reaction within the last 4 days or anaphylaxis within last month before planned ILIT or SCIT injection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-related immune cells in the FNA sample | At 2, 6 or 24 hours post allergen injection.
  An FNA of an inguinal lymph node will be performed at either 2, 6 or 24 hours after allergen injection depending on the individual randomization. The lymph node tissue will be evaluated for changes in cellular composition by mass cytometry (CyTOF). Multiple measurements (ca. 30) will be aggregated and described in a heat map.
Frequency of treatment-related immune cells in the blood samples sample | First bleeding on day 0. Second bleeding at 2, 6 or 24 hours post allergen injection. Third and fourth bleeding on days 7 and 28.
  Venous blood will be collected at first at baseline (day 0), then 2, 6 or 24 hours after allergen injection depending on the randomization, the on days 7 and 28 post allergen injection. The blood will be analysed by measuring cellular composition in whole blood by mass cytometry (CyTOF). Multiple measurements (ca. 30) will be aggregated and described in a heat map.

SECONDARY OUTCOMES:
Concentration of allergen-specific antibodies as a function of treatment | Day 0, day 7 and day 28.
  Allergen-specific antibodies will be measured as Units/ml in blood collected at baseline and after 7 and 28 days.
Concentration of leucocytes as a function of treatment | Day 0. Then 2, 4 or 24 hours post allergen injection. Then on days 7 and 28.
  A differential white blood cell count in blood collected at baseline and after 2, 4 or 24 hours, or after 7 and 28 days upon treatment will be measured using routine hematological diagnostics. The cell count will be quantified as number of cells per ml blood.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid-Grendelmeier, Prof. MD, Principal Investigator — University Hospital Zurich, Dept. Dermatology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD are coded for analysis. If data is to be shared with other researchers, the data will be coded.

REFERENCES:
- [Background] Aini NR, Mohd Noor N, Md Daud MK, Wise SK, Abdullah B. Efficacy and safety of intralymphatic immunotherapy in allergic rhinitis: A systematic review and meta-analysis. Clin Transl Allergy. 2021 Aug 17;11(6):e12055. doi: 10.1002/clt2.12055. eCollection 2021 Aug. PMID 34429875
- [Background] Jiang S, Xie S, Tang Q, Zhang H, Xie Z, Zhang J, Jiang W. Evaluation of Intralymphatic Immunotherapy in Allergic Rhinitis Patients: A Systematic Review and Meta-analysis. Mediators Inflamm. 2023 May 8;2023:9377518. doi: 10.1155/2023/9377518. eCollection 2023. PMID 37197570
- [Background] Werner MT, Bosso JV. Intralymphatic immunotherapy for allergic rhinitis: A systematic review and meta-analysis. Allergy Asthma Proc. 2021 Jul 1;42(4):283-292. doi: 10.2500/aap.2021.42.210028. PMID 34187620
- [Background] Hoang MP, Seresirikachorn K, Chitsuthipakorn W, Snidvongs K. Intralymphatic immunotherapy for allergic rhinoconjunctivitis: a systematic review and meta-analysis. Rhinology. 2021 Jun 1;59(3):236-244. doi: 10.4193/Rhin20.572. PMID 33647073
- [Background] Heath MD, Mohsen MO, de Kam PJ, Carreno Velazquez TL, Hewings SJ, Kramer MF, Kundig TM, Bachmann MF, Skinner MA. Shaping Modern Vaccines: Adjuvant Systems Using MicroCrystalline Tyrosine (MCT(R)). Front Immunol. 2020 Nov 24;11:594911. doi: 10.3389/fimmu.2020.594911. eCollection 2020. PMID 33324411
- [Background] Senti G, Johansen P, Kundig TM. Intralymphatic immunotherapy: from the rationale to human applications. Curr Top Microbiol Immunol. 2011;352:71-84. doi: 10.1007/82_2011_133. PMID 21725898
- [Result] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Result] Skaarup SH, Schmid JM, Skjold T, Graumann O, Hoffmann HJ. Intralymphatic immunotherapy improves grass pollen allergic rhinoconjunctivitis: A 3-year randomized placebo-controlled trial. J Allergy Clin Immunol. 2021 Mar;147(3):1011-1019. doi: 10.1016/j.jaci.2020.07.002. Epub 2020 Jul 15. PMID 32679209
- [Result] Skaarup SH, Graumann O, Schmid J, Bjerrum AS, Skjold T, Hoffmann HJ. The number of successful injections associates with improved clinical effect in intralymphatic immunotherapy. Allergy. 2021 Jun;76(6):1859-1861. doi: 10.1111/all.14642. Epub 2020 Nov 16. No abstract available. PMID 33099797

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT05960266/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT05960266/ICF_001.pdf